CLINICAL TRIAL: NCT02625012
Title: Repigmentation Patterns Induced by NB-UVB and Their Relationship With Melanocytic Dynamics in Vitiligo
Brief Title: Repigmentation Patterns Induced by NB-UVB and Their Relationship With Melanocytic Migration in Vitiligo
Acronym: UVBVIT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Juan Pablo Castanedo-Cazares (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Sponsor-Investigator, Juan Pablo Castanedo-Cazares, Clinical and research professor in Dermatology, Universidad Autonoma de San Luis Potosí
Organization: Universidad Autonoma de San Luis Potosí (Other)
Other Study IDs: UVVIT01
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Vitiligo
Keywords: Ultraviolet Therapy; Vitiligo; Melanocytes; Pigmentation
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vitiligo: A serial of vitiligo patients under treatment with UVB-NB

SUMMARY:
Vitiligo is the most common acquired depigmented disorder of the skin characterized by destruction of melanocytes resulting in well-circumscribed achromic macules. Ultraviolet phototherapy with narrow band (UVB-NB) is currently one of the treatments of choice, because it is able to induce proliferation, differentiation, maturation and migration of melanocytes. This repigmentation has distinctive patterns such as follicular, marginal, and diffuse. The aim of this study is to observe the dynamics of migration and proliferation, in vitiligo patients under UVB radiation phototherapy treatment. The investigators will evaluate this process by measuring FAK (focal adhesion kinase ) and c-Kit by immunohistochemistry and reverse transcriptase polymerase chain reaction assay.

DETAILED DESCRIPTION:
Vitiligo is the most common acquired depigmented disorder of the skin characterized by destruction of melanocytes, which results in well-circumscribed achromic macules. Its etiology is not fully recognized but functional melanocytes may disappear by autoimmune response, oxidative stress that induces melanocytes apoptosis, and loss of cell-cell adhesion between melanocytes and keratinocytes.

Ultraviolet phototherapy with narrow band (UVB-NB) is currently one of the treatments of choice with an average response rate of 60-70% on lesions. UVB-NB phototherapy may induce immune regulation and melanogenic induction. It is also able to induce Treg cells proliferation to suppress the autoimmune response which destroys melanocytes. By the other hand, UVB-NB induces signaling of proliferation, differentiation, maturation and migration of melanocytes, playing an important role in vitiligo re-pigmentation.

Phosphorylation of focal adhesion kinase (p-FAK125) is a cytoplasmic tyrosine kinase that plays as an important component in the signal transduction of cell migration, as it modulates cytoskeletal proteins necessary for their movement. UVB-NB radiation induces migration on melanocytes cultures increasing their levels of p-FAK125 and it has been proposed as a melanocyte migration marker.

C-kit is a tyrosine kinase receptor expressed on melanoblasts and differentiated melanocytes. Ligand binding induces PI3K, MAPK and Src kinase pathways, which traduce differentiation of melanoblast into proliferating melanocytes; so its expression imply the presence of mature pigmented melanocytes. C-kit is increased in mature melanocytes after UVB exposure, but it has been show that in melanoma cases the loss of c-kit expression is involved in cancer progression , therefore c-kit signaling is also associated in migratory process. Although, different reports have been established the expression of this markers on vitiligo, is not defined this markers on the repigmentation patterns induces to UVB radiation.

UVB radiation induces repigmentation in distinctive patterns such as follicular, marginal, and diffuse. Follicular pattern is the predominant, and comes from hair follicle melanocytes. In the marginal pattern melanocytes from healthy skin are attracted to the lesion. In the diffuse pattern UVB radiation stimulates those inactive melanocytes. In contrast, achromic pattern not induces melanocyte activation. The relation between the biological behavior of melanocytes and these repigmentation patterns, may provide insights to an improved method to treat vitiligo. The aim of this study is to observe the dynamic of migration and proliferation by specific markers on the repigmentation patterns of vitiligo patients under UVB radiation phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* Symmetric vitiligo
* Affected body surface greater than 15%
* Patients with follicular, marginal and diffuse repigmenting patterns
* No previous topical or systemic treatment
* Signed informed consent

Exclusion Criteria:

* Concomitant treatment or systemic diseases
* Pregnancy
* Drugs intake
* Mental disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical diagnosis of vitiligo vulgaris
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Melanocyte phenotype | Up to 1 year
  To quantify melanocyte maturation stages in vitiliginous skin through markers

SECONDARY OUTCOMES:
Melanocyte number | Up to 1 year
  To quantify the number of melanocytes in vitiliginous skin lesions
Melanogenesis characteristics | Up to 1 year
  To quantify the expression of melanogenic in vitiliginous skin lesions
Melanin presence | Up to 1 year
  To quantify melanin epidermal deposition in vitiliginous skin lesions

CONTACTS AND LOCATIONS:
Overall Officials: Diego Cortes-Garcia, PhD, Principal Investigator — Universidad Autonoma de San Luis Potosi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lepe V, Moncada B, Castanedo-Cazares JP, Torres-Alvarez MB, Ortiz CA, Torres-Rubalcava AB. A double-blind randomized trial of 0.1% tacrolimus vs 0.05% clobetasol for the treatment of childhood vitiligo. Arch Dermatol. 2003 May;139(5):581-5. doi: 10.1001/archderm.139.5.581. PMID 12756094
- [Background] Castanedo-Cazares JP, Lepe V, Moncada B. Repigmentation of chronic vitiligo lesions by following tacrolimus plus ultraviolet-B-narrow-band. Photodermatol Photoimmunol Photomed. 2003 Feb;19(1):35-6. doi: 10.1034/j.1600-0781.2003.00005.x. No abstract available. PMID 12713553
- [Background] Picardo M, Bastonini E. A New View of Vitiligo: Looking at Normal-Appearing Skin. J Invest Dermatol. 2015 Jul;135(7):1713-1714. doi: 10.1038/jid.2015.92. PMID 26066890
- [Background] Wu CS, Lan CC, Yu HS. Narrow-band UVB irradiation stimulates the migration and functional development of vitiligo-IgG antibodies-treated pigment cells. J Eur Acad Dermatol Venereol. 2012 Apr;26(4):456-64. doi: 10.1111/j.1468-3083.2011.04094.x. Epub 2011 May 4. PMID 21545543